CLINICAL TRIAL: NCT01160302
Title: An Exploratory Biomarker Trial of the Food Substances Curcumin C3 Complex® in Subjects With Newly Diagnosed Head and Neck Squamous Cell Carcinoma
Brief Title: Curcumin Biomarker Trial in Head and Neck Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Collaborators: Feist-Weiller Cancer Center at Louisiana State University Health Sciences (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Cherie Ann Nathan, Chairman, Dept of Otolaryngology, Louisiana State University Health Sciences Center Shreveport
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H08-081; 1R21CA137545-01A2 (NIH); FWCC (Other: Feist-Weiller Cancer Center)
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Head and Neck Cancer
Keywords: cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Microgranular Curcumin (Experimental): Consume 4g microgranular curcumin (Curcumin C3 Complex) twice per day
  Interventions: Drug: Microgranular Curcumin C3 Complex®

INTERVENTIONS:
Drug: Microgranular Curcumin C3 Complex® — 4 grams twice daily for 21-28 days

SUMMARY:
There is considerable evidence that turmeric consumption may have a protective effect against cancer progression. The purpose of this study is to examine the short-term effects of supplementation with a turmeric extract, Curcumin C3 Complex®, on biomarkers of head and neck squamous cell carcinoma (HNSCC).

DETAILED DESCRIPTION:
This is an open label, exploratory biomarker trial of the food substances Curcumin C3 Complex® in subjects with newly diagnosed HNSCC. Curcumin, a novel safe nutritional interventional agent has exciting potential usage as a preventive/adjuvant agent, and prevents tumor formation by inhibiting an important molecular pathway that is shown to cause cancer progression, which we will test as a tumor marker in this clinical trial.

The primary objective is to evaluate biomarker response of HNSCC patients to the food substances Curcumin C3 Complex®. This will be done by comparing post-intervention values to baseline values. In addition, we will determine the levels of curcumin and its metabolites in tumor and adjacent tissue.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with newly diagnosed head and neck squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx and have at least one accessible tumor
* Subjects willing to undergo tumor biopsies
* Subjects willing to refrain from nonsteroidal anti-inflammatory drugs (NSAIDS)
* Eastern Co-operative Oncology Group (ECOG) status of 0-3
* Absolute Neutrophil Count ≥ 1500/mm³, Hgb ≥ 10g/dl and Platelet count ≥ 150,000 mm3
* Adequate Renal Function: serum creatinine ≤ 1.5 × upper limit of normal (ULN). Adequate hepatic function: total bilirubin ≤ 1.5 × ULN, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.0 × ULN
* Signed and dated institutional review board approved informed consent form before any protocol specific procedures are performed
* Willingness of subjects who are not surgically sterile or postmenopausal to use reliable methods of birth control for the duration of the study and for 2 weeks after last dose of study drug
* No consumption of curcumin-rich foods to subject's knowledge within the previous 48 hours
* Age ≥ 18 years to ≤ 90 years

Exclusion Criteria:

* Subjects receiving anticoagulation therapy
* Known hypersensitivity to curry or black pepper
* Prior cancer therapy in the last 30 day
* Concurrent chemotherapy or radiation
* Severely immunocompromised subjects
* Subjects known to be HIV positive
* any major illness that, in the investigator's judgment, will substantially increase the risk asociated with the subject's participation in the study
* Pregnant or nursing women
* Unwillingness or inability to comply with required study visits and procedures in this protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in tissue biomarkers | 21-28 days
  Change in tissue levels, between pre- and post-treatment biopsy
Pharmacokinetics of microgranular curcumin | 21-28 days
  Determine whether biologically active levels of curcumin can be achieved in head and neck tumors

SECONDARY OUTCOMES:
Ease of ingestion | 21-28 days
  Determine if microgranular curcumin can be easily ingested

CONTACTS AND LOCATIONS:
Overall Officials: Cherie-Ann O Nathan, MD, FACS, Principal Investigator — LSUHSC-Shreveport and Feist-Weiller Cancer Center
Locations (1):
- LSUHSC-Shreveport and Feist-Weiller Cancer Center, Shreveport, Louisiana, United States